CLINICAL TRIAL: NCT00267514
Title: A Randomized, Cross-over Study to Demonstrate Equivalence of Sevelamer Carbonate Powder and Sevelamer Hydrochloride Tablets Dosed Three Times Per Day in Haemodialysis Patients
Brief Title: Study to Demonstrate Equivalence of Sevelamer Carbonate Powder and Sevelamer HCl Tablets in Haemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SVCARB00205
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

ARMS (2):
- 1 (Other): sevelamer carbonate powder x 4 weeks then, sevelamer hydrochloride x 4 weeks
  Interventions: Drug: sevelamer carbonate (Renvela®) sevelamer hydrochloride (Renagel ®)
- 2 (Other): sevelamer hydrochloride x 4 weeks then, sevelamer carbonate powder x 4 weeks
  Interventions: Drug: sevelamer hydrochloride (Renagel ®) sevelamer carbonate (Renvela®)

INTERVENTIONS:
Drug: sevelamer carbonate (Renvela®) sevelamer hydrochloride (Renagel ®) — sevelamer carbonate powder dosed TID with meals for four weeks followed by sevelamer hydrochloride tablets dosed TID with meals for four weeks
  Arms: 1
Drug: sevelamer hydrochloride (Renagel ®) sevelamer carbonate (Renvela®) — sevelamer hydrochloride tablets dosed TID with meals for four weeks followed by sevelamer carbonate powder dosed TID with meals for four weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine if sevelamer carbonate powder is an effective treatment for the control of serum phosphorous levels in patients on dialysis when compared to sevelamer hydrochloride tablets.

ELIGIBILITY:
Inclusion Criteria:

* Receiving three times per week haemodialysis for three months or longer.
* Taking sevelamer hydrochloride alone (e.g. not using other types of phosphate binders concomitantly) or on combination therapy (e.g. using sevelamer hydrochloride and calcium containing, or metal phosphate binders concomitantly) not exceeding a total daily binder dose of 14.4 g, for at least 60 days prior to screening.
* Have the following documented local laboratory measurements:

  1. Two most recent consecutive serum phosphorus measurements that are ≥ 3.0 and ≤ 7.0 mg/dL (≥ 0.96 and ≤ 2.26 mmol/L) within 60 days of screening
  2. An most recent iPTH measurement ≤ 900 pg/mL (< 99 pmol/L) within 90 days of screening
  3. A most recent serum calcium (adjusted for albumin) measurement within normal range defined by the local laboratory within 60 days of screening
* Have the following central laboratory measurements:

  1. A serum phosphorus measurement ≥ 5.5 mg/dL (≥ 1.76 mmol/L) at Visit 2 (after Washout)
  2. A serum iPTH measurement ≤ 800 pg/mL at Visit 5 (prior to randomization)
  3. A serum phosphorus measurement ≥ 3.0 and ≤ 6.5 mg/dL (≥ 0.96 and ≤ 2.08 mmol/L) at Visit 5
* If on vitamin D replacement or calcimimetics therapy, be at a stable dose for at least one month prior to screening and willing to maintain the same dose throughout the duration of the study, except for safety reasons.
* Willing to maintain screening doses of lipid medication for the duration of the study, except for safety reasons.
* Willing to avoid any intentional changes in diet such as fasting or dieting.
* If female and of childbearing potential (pre-menopausal and not surgically sterile), willing to use an effective contraceptive method throughout study, which includes barrier methods, hormones, or intrauterine devices (IUDs).
* Willing to stop all calcium supplements not prescribed by the investigator including multivitamins containing calcium.
* Willing to refrain from using aluminium, calcium, lanthanum, or magnesium containing antacids throughout duration of the study unless prescribed by the investigator as a calcium supplement per protocol.
* Have a level of understanding and willingness to cooperate with all visits and procedures, including telephone contacts, as described in the consent by the study site personnel.

Exclusion Criteria:

* Have poorly controlled diabetes mellitus or hypertension, active vasculitis, HIV infection, or any clinically significant unstable medical condition (defined by investigator).
* Have active dysphagia, swallowing disorders, bowel obstruction, or severe gastrointestinal motility disorders.
* Have participated in a study of an investigational drug during the 30 days preceding the start of the screening period.
* Has active ethanol or drug dependence or abuse, excluding tobacco use.
* Have any other condition, which, in the investigator's opinion, will prohibit the patient's participation in the study.
* If female, be pregnant or breast-feeding.
* Have any evidence of active malignancy except for basal cell carcinoma of the skin. A history of malignancy is not an exclusion.
* Use of anti-arrhythmic or anti-seizure medications for arrhythmia or seizure disorders.
* Have a known hypersensitivity to sevelamer or any of its constituents.
* Have a poor record of compliance with medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Demonstrate the equivalence of sevelamer carbonate powder to sevelamer hydrochloride tablets dosed three times per day (TID) with meals on the control of serum phosphorus levels | Up to 13 weeks
Evaluate the safety and tolerability of sevelamer carbonate powder compared to sevelamer hydrochloride tablets dosed TID with meals | Up to 13 weeks

SECONDARY OUTCOMES:
Compare the effects of sevelamer carbonate powder to sevelamer hydrochloride tablets when dosed three times a day with meals on: serum calcium-phosphorus product | Up to 13 weeks
serum lipid profile (total cholesterol, high density lipoprotein [HDL] and low density lipoprotein [LDL] and triglycerides) | Up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- United Kingdom (7):
  - Southmead Hospital, Bristol
  - Addenbrooks NHS Trust, Cambridge
  - The Royal London Hospital, London
  - Guy's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Hope Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich